CLINICAL TRIAL: NCT02051023
Title: Randomized, Double-Masked, Vehicle-controlled Phase III Trial on the Safety/Efficacy of FML® 0.1% in the Treatment of the Inflammatory Exacerbation Provoked by Exposure to an Adverse Controlled Environment in Patients With Dry Eye Disease
Brief Title: Efficacy and Safety of Fluorometholone (FML) in Dry Eye Disease (Keratoconjunctivitis Sicca)
Acronym: FML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IOBA-CERLAB-003-2013
Record Dates: First submitted 2014-01-22; First posted 2014-01-31 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Dry Eye
Keywords: keratoconjunctivitis sicca; dry eye; dry eye syndrome; dry eye disease; steroids
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — Fluorometholone; Ophthalmic Solutions; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FML 0.1% eyedrops (Experimental): FML (fluorometholone) 0.1% eyedrops 4 times a day in both eyes for 22 days
  Interventions: Drug: FML 0.1% eyedrops
- Liquifilm artificial tears eyedrops (Active Comparator): Topical application 4 times a day in both eyes for 22 days
  Interventions: Drug: Liquifilm artificial tears eyedrops

INTERVENTIONS:
Drug: FML 0.1% eyedrops — Ocular topical application of fluorometholone 0.1% 4 times a day during 22 days
  Other Names: 0.1% fluorometholone
  Arms: FML 0.1% eyedrops
Drug: Liquifilm artificial tears eyedrops — Liquifilm instillation 4 times a day for 22 days
  Other Names: Artificial tears
  Arms: Liquifilm artificial tears eyedrops

SUMMARY:
Hypothesis: Fluorometholone (FML) 0.1% eyedrops topically applied 4 times a day for 22 days is more efficient than artificial tears (Liquifilm) in dry eye disease (DED) and ameliorates the worsening of the disease after exposure to an adverse controlled environment.

DETAILED DESCRIPTION:
There will be 4 visits in 3 different days:

Visit 1 (V1). Inclusion in normalized controlled environment (NCE)

Visit 2 (V2). 21 days post-treatment. Data collected in NCE

Visit 3 (V3). 21 days post-treatment. Data collected in adverse controlled environment (ACE)

Visit 4 (V4). 22 days post-treatment. Recovery visit in ACE. Data collected in NCE

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Signed informed consent
* Subjects refer worsening in their pathologies when exposed to adverse environmental conditions in their daily life
* Fluorescein corneal staining ≥ 1in Oxford Scale
* Ocular surface disease index (OSDI) test > 12
* Tear breakup Time (TBT) ≤ 7 seconds in both eyes
* Schirmer test without anesthesia ≤ 10 mm in 5 minutes in both eyes
* Any concomitant medication that may affect dry eye syndrome, ocular surface or vision, must have started at least 3 months before screening visit, and there are no changes in dose expected during the study duration.
* Best corrected visual acuity at least 0.1 logMar at 6 meters with both eyes
* Current use of ophthalmic artificial tears at study inclusion.
* Signed informed consent
* Signed data protection consent

Exclusion Criteria:

* Sensitivity or known intolerance to any of the products used in the study
* Previous severe ocular inflammation or infections in the 6 previous months to study inclusion
* Any ocular pathology other than dry eye syndrome or atopic keratoconjunctivitis
* Any ocular surgery or trauma that may affect corneal sensitivity and / or normal tear distribution (refractive or cataract surgery) in the 6 previous months or any ocular or systemic surgery planned during the study duration that may affect the study as assessed by principal investigator.
* Use of contact lenses in the 3 previous months to study inclusion
* Use of any topical medication for pathologies other than dry eye syndrome.
* Any ocular topical treatment for dry eye syndrome with corticosteroids or non steroid anti-inflammatory drugs must have stopped 1 month before study inclusion. Any treatment with topical cyclosporin must have been stopped 3 months before study inclusion.
* Any uncontrolled severe systemic disease that may affect the eye (except for Sjögren Syndrome)
* Start, discontinuation or dose change during the study of antihistaminic, cholinergic agents, beta blockers, antidepressants or any other systemic medications with potential effect over tear film.
* Start of any systemic treatment that may affect dry eye syndrome, vision, ocular surface or intraocular pressure during the 3 previous months to study inclusion.
* Surgical / non surgical tear point occlusion in the 3 previous months to study inclusion or prevision during study duration for this procedure.
* Cup / disc ratio > 0.6
* History of intraocular pressure > 22 mm Hg within 2 months previous to study inclusion
* Pregnancy or breastfeeding women
* Inclusion in another research study in the previous 30 days to study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Fluorescein corneal staining | 22 days
  Evidence of statistically significant changes in the number of subjects with an increase ≥ 1 point in fluorescein corneal staining between pre and post adverse condition exposure in ACE (V2 vs V3) and between post adverse condition exposure in ACE and recovery visit (V3 vs V4).
Symptom Assessment in Dry Eye (SANDE) I and II questionnaire | 22 days
  Evidence of statistically significant changes in the number of subjects with a reduction ≥ 2 points in SANDE score between pre and post adverse condition exposure in ACE (V2 vs V3) and between post adverse condition exposure and recovery visit (V3 vs V4).

SECONDARY OUTCOMES:
Tear inflammatory molecule levels | 22 days
  Evidence of statistically significant changes between the differences in tear molecule concentrations pre and post adverse condition exposure (V2 vs V3) in ACE and between post adverse condition exposure and recovery visit (V3 vs V4).
Best corrected visual acuity | 22 days
  Best corrected visual acuity measured with the ETDRS (Eearly Treatment for Diabetes Retinopathy Study) chart after 22 days of treatment compared to baseline
Biomicroscopy findings at slit lamp examination | 22 days
  Biomicroscopy findings (general aspect of ocular surface and anterior segment, plus corneal and conjunctival staining) after 22 days of treatment compared to baseline
Adverse events during the trial | 22 days
  Adverse events that occur during the trial
Other Efficacy Measures | 22 days
  Conjunctival Staining (Lissamine Green; Oxford Scale) T-BUT (tear break-up time) Conjunctival hyperemia (Efron Scale) Patient satisfaction with the treatment (VAS 0-100)
Intraocular pressure (IOP) and fundus examination | 22 days
  Intraocular pressure levels measured with a Goldman tonometer Evaluation of optic disk/cup ratio at fundus examination

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Calonge-Cano, MD, PhD, Principal Investigator — Ocular surface group Director - IOBA
Locations (2):
- Spain (2):
  - IOBA (Instituto de Oftalmobiología Aplicada), University of Valladolid, Valladolid, Valladolid
  - IOBA, Valladolid, Valladolid